CLINICAL TRIAL: NCT00472147
Title: Selection of Shock Energy in Out-Of-Hospital Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBF-2007002
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2007-05-11 (Estimated); Status verified 2007-05

CONDITIONS: Sudden Cardiac Death; Arrhythmia; Survival
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: shock efficacy

SUMMARY:
Sudden cardiac death is the most frequent cause of death in industrialized countries. The most efficient interventiont in ventricular fibrillation is defibrillation in an appropriate timely manner. But since the intervention of defibrillation the optimal shock energy is unknown. As a too low energy is not able to terminate ventricular fibrillation a too high energy may cause asystole wich jeopardizes survival itself. We study the efficacy of different shock energies on the termination of ventricular fibrillatiion and survival.

ELIGIBILITY:
Inclusion Criteria:

* out of hospital sudden cardiac death
* ventricular fibrillation

Exclusion Criteria:

* non cardiac death
* asystole

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
termination of vf survival

SECONDARY OUTCOMES:
resulting rhythm CPC score

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Müller, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité campus Benjamin Franklin, Berlin, State of Berlin, Germany